CLINICAL TRIAL: NCT05809921
Title: Dual IntraVenous Thrombolysis Approach (DIVA) in Patients With Medium-vessel-occlusion Strokes: a Retrospective Study
Acronym: DIVArétro
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0002
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke Due to Medium-vessel-occlusion
Keywords: Acute stroke; Medium-vessel occlusion; Thrombolysis; Tenecteplase
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single-IVT strategy (SIS) cohort: The SIS cohort included patients with MeVO strokes who received a single conventional alteplase IVT (IVT-1).
  Interventions: Drug: alteplase
- Dual-IVT strategy (DIS) cohort: The DIS cohort included patients with alteplase-treated MeVO strokes for whom a repeat MRI (MRI-2) was planned 1-2h after alteplase IVT (IVT-1) to discuss a possible complementary IVT with tenecteplase (TNK-IVT-2).
  Patients could be in the following situations: already recanalized at 1-2h post-alteplase IVT-1, persistent occlusion treated with TNK-IVT-2 or persistent occlusion but additional IVT contraindicated according to the study protocol.
  Interventions: Drug: Alteplase + possible complementary IVT with tenecteplase

INTERVENTIONS:
Drug: alteplase — Intravenous thrombolysis with alteplase (0.9 mg/kg, maximum 90 mg) with 10% of the dose given as a bolus followed by an infusion lasting 60 minutes.
  Groups: Single-IVT strategy (SIS) cohort
Drug: Alteplase + possible complementary IVT with tenecteplase — Intravenous thrombolysis with alteplase (0.9 mg/kg, maximum 90 mg, with 10% of the dose given as a bolus followed by an infusion lasting 60 minutes) and depending on the MRI-2 results, an additional IVT with tenecteplase (0.25mg/kg, maximum 25 mg, with 100% of the dose given as a bolus) could be given in case of persistent occlusion and with no contraindication according to the study protocol.
  Groups: Dual-IVT strategy (DIS) cohort

SUMMARY:
The purpose of this study (Dual IV thrombolysis Approach (DIVA) study) is to assess a new medical strategy for Medium-vessel-occlusion (MeVO) strokes, based on a second IV thrombolysis with tenecteplase (TNK) for persistent intracranial occlusion on MRI 1-2 hours after standard alteplase infusion. The DIVA-study results were compared with a similar cohort of MeVO strokes patients treated with standard therapy (single IVT with alteplase) during the same timeframe in another stroke unit.

DETAILED DESCRIPTION:
MeVO strokes account for 25-40% of all acute ischemic stroke (AIS). In a recent study, less than 1/3 of MeVO strokes patients had a so-called "minor stroke" (National Institute of Health Stroke score (NIHSS)<6), thereby emphasizing that strategically located MeVO strokes can be debilitating. Therefore it is crucial to achieve early recanalization, which is strongly associated with excellent outcomes. However, standard medical treatment (that is to say, a single intravenous thrombolysis (IVT) with alteplase 0.9mg/kg) resulted in early (60-120 min) and late (24-36 hours) recanalizations of MeVO in only 30% and 64% respectively. As a consequence, and in line with a recent study, almost 40% of these patients were functionally dependent at 3 months (modified Rankin Score>2) despite IVT.

Because randomized clinical trials on EVT enrolled only limited numbers of patients with distal occlusions, mostly proximal M2 segment-middle cerebral artery occlusions, EVT has not yet been established as standard-of-care for MeVO strokes, and owing to the fragility of these small intracranial arteries, safety of EVT for MeVO is questionable and randomized trials are ongoing.

In comparison with EVT, a purely chemical strategy for MeVO strokes would be far less human-resource demanding, cheaper and feasible almost everywhere. In a previous study, the investigators showed results in favor of a high rate of recanalization at 24h in patients with stroke due to proximal occlusion with a dual IVT strategy (additional IVT with TNK in patients with persistent occlusion 1h after alteplase IVT), and this with a low hemorrhagic risk. Distal arterial occlusions are at lower hemorrhagic risk than proximal occlusions because volume infarcts are smaller, and because they spare basal ganglia, a critical location for massive hemorrhagic transformation of AIS. Moreover, patients could be carefully pre-selected with the initial MRI evaluation, allowing exclusion of patients with severe microangiopathy or amyloid angiopathy.

From March 1, 2014, to November 31, 2018, the investigators proposed a dual-IVT strategy (DIS) to patients admitted to the CHSF-Stroke Unit for MeVO-associated AIS eligible for IVT but not suitable for EVT. They were given a repeat MRI 1-2h after alteplase, 0.9 mg/kg, maximum 90 mg (IVT-1). If no recanalization was obtained and in the absence of exclusion criteria (acute lesion visible on FLAIR sequence, new cerebral/subarachnoid hemorrhage; significant extracerebral bleeding), a second IVT with TNK, 0.25 mg/kg, maximum 25 mg) (IVT-2) was given. The whole procedure was done within 6h of symptom onset.

During the same period, Bordeaux University Hospital-Stroke Unit constituted a cohort of consecutive patients with MeVO-AIS treated with conventional single-IVT strategy (SIS) using alteplase.

DIS- and SIS-cohort data were collected prospectively and the comparison was retrospective.

The pre-specified primary efficacy endpoint was successful recanalization assessed on MRI at 24h. The pre-specified primary safety endpoint was severe bleeding: symptomatic intracranial hemorrhage or major systemic bleeding during the first 36 hours. Secondary endpoints were: early neurological improvement at 24h, early complete neurological recovery at 24h and excellent (modified Rankin scale (mRS) 0-1) and good (mRS 0-2) clinical outcomes at 3 months.

ELIGIBILITY:
Inclusion Criteria:

For the SIS cohort :

* Age≥ 18 years
* Acute ischemic stroke (visible on DWI, but not visible on FLAIR) on initial MRI associated with distal arterial occlusion as defined below:

  * A distal occlusion of the M2 segment of the middle cerebral artery (MCA)
  * Occlusion (regardless of location) of a non-dominant M2 branch of the MCA
  * Occlusion of the M3 segment of the MCA.
  * Occlusion of the A2 or A3 segment of the anterior cerebral artery (ACA)
  * Occlusion of the P2 or P3 branch of the posterior cerebral artery (PCA).
  * A proximal M2-MCA or proximal P1-PCA occlusion may also be included if not eligible for mechanical thrombectomy, especially if the initial NIHSS score is low (<5).
* IVT by ALT within 4h30 after onset of symptoms,
* MRI performed 24h after IVT

For the DIS cohort :

* Age≥ 18 years
* Acute ischemic stroke (visible on DWI, but not visible on FLAIR) on baseline MRI associated with distal arterial occlusion as defined below:

  * A distal occlusion of the M2 segment of the middle cerebral artery (MCA)
  * Occlusion (regardless of location) of a non-dominant M2 branch of the MCA
  * Occlusion of the M3 segment of the MCA.
  * Occlusion of the A2 or A3 segment of the anterior cerebral artery (ACA)
  * Occlusion of the P2 or P3 branch of the posterior cerebral artery (PCA).
  * A proximal M2-MCA or proximal P1-PCA occlusion may also be included if not eligible for mechanical thrombectomy, especially if the initial NIHSS score is low (<6).
* IVT by ALT within 4h30 after onset of symptoms
* Repeat MRI performed 1-2h after IVT (MRI-2)
* Brain MRI performed 24h after IVT

Exclusion Criteria:

Inclusion Criteria:

For the SIS cohort :

* Age≥ 18 years
* Acute ischemic stroke (visible on DWI, but not visible on FLAIR) on initial MRI associated with distal arterial occlusion as defined below:

  * A distal occlusion of the M2 segment of the middle cerebral artery (MCA)
  * Occlusion (regardless of location) of a non-dominant M2 branch of the MCA
  * Occlusion of the M3 segment of the MCA.
  * Occlusion of the A2 or A3 segment of the anterior cerebral artery (ACA)
  * Occlusion of the P2 or P3 branch of the posterior cerebral artery (PCA).
  * A proximal M2-MCA or proximal P1-PCA occlusion may also be included if not eligible for mechanical thrombectomy, especially if the initial NIHSS score is low (<5).
* IVT by ALT within 4h30 after onset of symptoms,
* MRI performed 24h after IVT

For the DIS cohort :

* Age≥ 18 years
* Acute ischemic stroke (visible on DWI, but not visible on FLAIR) on baseline MRI associated with distal arterial occlusion as defined below:

  * A distal occlusion of the M2 segment of the middle cerebral artery (MCA)
  * Occlusion (regardless of location) of a non-dominant M2 branch of the MCA
  * Occlusion of the M3 segment of the MCA.
  * Occlusion of the A2 or A3 segment of the anterior cerebral artery (ACA)
  * Occlusion of the P2 or P3 branch of the posterior cerebral artery (PCA).
  * A proximal M2-MCA or proximal P1-PCA occlusion may also be included if not eligible for mechanical thrombectomy, especially if the initial NIHSS score is low (<6).
* IVT by ALT within 4h30 after onset of symptoms
* Repeat MRI performed 1-2h after IVT (MRI-2)
* Brain MRI performed 24h after IVT

Exclusion Criteria

For SIS and DIS cohort :

* Patients informed of the study who objected to the collection of their data.
* Patients with >5 microbleeds; diffuse or focal cortical siderosis; severe leukoaraiosis (Fazekas score 3/3); any coagulopathy type, including a baseline international normalized ratio (INR) >1.3, were excluded for the SIS and DIS cohort.

Exclusion criteria for a complementary IVT with TNK in the DIS cohort:

(Patients will be included in the DIS cohort but will not receive a secondary IVT with TNK ) Brain exclusion criteria on MRI-2: Early recanalization, acute lesion visible on FLAIR sequence, new cerebral/subarachnoid hemorrhage of any type or size.

Significant extracerebral bleeding, such as abundant gingivorrhagia, epistaxis, multiple/diffuse ecchymoses or macroscopic hematuria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a bicentric retrospective study: Sud-Francilien Hospital (SFH), Corbeil-Essonnes, France for the DIVA cohort and Bordeaux University Hospital (BUH) for the standard treatment with alteplase alone cohort, based on stroke registries prospectively gathered.
  From March 2014 to November 2018, consecutive patients in SFH and BUH with acute ischemic stroke (AIS) due to distal occlusion assessed on brain MRI who fulfilled the inclusion/exclusion criteria were included in this retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Recanalization rate assed on the control MRI at 24h (MRI-3) based on the Arterial Occlusive Lesion (AOL) score | at 24 hours
  Recanalization rate at 24h was evaluated on MRI-3 using the AOL scale. This scale was adapted for very distal occlusions which are not always clearly visible on magnetic resonance angiography (MRA). In these cases, AOL scale-score was based on gradient echo-sequences (GE):
  If occlusion visible on MRI:
  * no recanalization: AOL- 0, 1, 2a
  * successful recanalization : AOL-2b or 3
  If occlusion not visible on MRA but thrombus visible on GE:
  * no recanalization : AOL-0 (unchanged thrombus) or AOL-1/AOL-2a (slight down-stream migration ore size reduction of the thrombus)
  * successful recanalization : AOL-2b (residual distal thrombus), or AOL-3 (complete thrombus disappearance).

SECONDARY OUTCOMES:
Symptomatic intracranial Hemorrhages (sICH) | at 24 hours
  Rates of sICH at 24h (on MRI-3) according to the SITS-MOST and ECASS II criteria.
NIHSS | at 24 hours
  Clinical severity based on NIHSS assessment Delta NIHSS : NIHSS-H0 minus NIHSS-H24 Based on NIHSS assessment : baseline, at 24h. Delta NIHSS : NIHSS-H0 minus NIHSS-H24
modified Rankin Scale score (mRS) | at 3 months
  Functional independency
mRS 6 | at 3 months
  death

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chausson N, Olindo S, Laborne FX, Aghasaryan M, Renou P, Soumah D, Debruxelles S, Altarcha T, Poli M, L'Hermitte Y, Sagnier S, Toudou-Daouda M, Aminou-Tassiou NR, Bentamra L, Benmoussa N, Alecu C, Imbernon C, Smadja L, Ouanounou G, Rouanet F, Sibon I, Smadja D. Second-dose intravenous thrombolysis with tenecteplase in alteplase-resistant medium-vessel-occlusion strokes: A retrospective and comparative study. Eur Stroke J. 2024 Dec;9(4):943-951. doi: 10.1177/23969873241254936. Epub 2024 Jun 3. PMID 38829011